CLINICAL TRIAL: NCT05365971
Title: RISE FOR HEALTH Study by the PLUS Consortium
Brief Title: RISE FOR HEALTH Study
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of California, San Diego (Other); University of Pennsylvania (Other); Yale University (Other); University of Michigan (Other); Loyola University Chicago (Other); University of Alabama at Birmingham (Other); Washington University School of Medicine (Other); Northwestern University (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00012315
Record Dates: First submitted 2022-04-28; First posted 2022-05-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Bladder Health; LUTS; PLUS; RISE
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and vaginal swab; additionally stool for subset
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The RISE FOR HEALTH study (RISE) is an initiative of the Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium, which was formed by the NIDDK in 2015 to develop the science to improve bladder health in women and girls. RISE is designed to identify risk and protective factors for bladder health and lower urinary tract symptoms (LUTS) and to estimate the distributions of bladder health and bladder health knowledge, attitudes, and beliefs in women of all ages across the life course.

This will be accomplished by conducting a population-based prospective cohort study. A sample of individuals who live within the study base, i.e., the county containing each PLUS clinical research center and each adjacent county, will be invited to complete two baseline surveys and then two follow-up surveys one year later. A subset of participants will be invited to attend an in-person evaluation to collect additional clinical information and biologic specimens.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* Age ≥18 years
* Identify or born as female (includes cis- and trans-women, and trans-men)
* Able to read and understand English or Spanish
* Able to read and provide informed consent

Exclusion Criteria:

* Physical or mental health conditions that would prohibit self-administration of questionnaires either electronically or using paper and pencil (e.g., dementia/cognitive impairment/blindness/severe arthritis).
* Residence in a nursing home or other institutionalized living facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female or have female listed on their birth certificate (including cisgender women, trans men, trans women, and non-binary persons)
Study Population: The source population for RISE will be adult (18 years of age or older) cis-gendered women, trans-men, and trans-women from the resident, civilian, non-institutionalized US population capable of completing a survey in English or Spanish (see eligibility criteria for exact criteria).
Sampling Method: Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Bladder Health Scales and Function Indices | Baseline assessment
  Multi-item measurement to assess bladder health comprised of subscales and indices ranging from zero to 100

SECONDARY OUTCOMES:
Knowledge, Attitudes and Beliefs (KAB) | Baseline assessment
  Several questions on knowledge, attitudes, and beliefs regarding bladder health and influences on bladder health
Change in Bladder Health Scales and Function Indices | 1 year follow-up from baseline assessment
  Change in multi-item measurement to assess bladder health comprised of subscales and indices ranging from zero to 100

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Sutcliffe, PhD, Study Chair — Washington University School of Medicine; Ariana Smith, MD, Study Chair — University of Pennsylvania
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Loyola University Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Submission to NIDDK central repository.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Smith AL, Sutcliffe S; Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium. Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium-Update for Society of Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction (SUFU). Neurourol Urodyn. 2026 Feb 4. doi: 10.1002/nau.70230. Online ahead of print. PMID 41640096